CLINICAL TRIAL: NCT03192644
Title: The Impact on Recurrence Risk of Adjuvant Transarterial Chemoinfusion (TAI) Versus Adjuvant Transarterial Chemoembolization (TACE) for Patients With Hepatocellular Carcinoma And Portal Vein Tumor Thrombosis (PVTT) After Hepatectomy : A Random, Controlled, Stage III Clinical Trial.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Rong-ping Guo, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2017-004-01
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Epirubicin; Cisplatin; Ethiodized Oil; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (TAI) (Experimental)
  Interventions: Procedure: TAI; Drug: mFOLFOX6 (oxaliplatin, calcium folinate, and 5-FU)
- Group B (TACE) (Active Comparator)
  Interventions: Procedure: TACE; Drug: epidoxorubicin and cisplatin and lipiodol

INTERVENTIONS:
Procedure: TAI — transarterial chemoinfusion with mFOLFOX6 (oxaliplatin, calcium folinate, and 5-FU)
  Arms: Group A (TAI)
Procedure: TACE — transarterial chemoembolization with epidoxorubicin and cisplatin and lipiodol
  Arms: Group B (TACE)
Drug: epidoxorubicin and cisplatin and lipiodol — epidoxorubicin and cisplatin and lipiodol
  Arms: Group B (TACE)
Drug: mFOLFOX6 (oxaliplatin, calcium folinate, and 5-FU) — oxaliplatin, calcium folinate, and 5-FU
  Arms: Group A (TAI)

SUMMARY:
To compare the impact on recurrence risk of adjuvant TAI and adjuvant TACE for patients with HCC and PVTT after hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old and younger than 75 years;
* ECOG PS<3;
* proven hepatocellular carcinoma with PVTT according pathological examination;
* not previous treated for tumor;
* tumor and tumor thrombosis were removed in operation;
* no recurrence occurence at 4 to 7 weeks after surgery;
* the lab test could meet: neutrophil count≥1.5×109/L; hemoglobin≥80g/L; platelet count≥60×109/L; serum albumin≥28g/L; total bilirubin<3-times upper limit of normal; ALT<5-times upper limit of normal; AST<5-times upper limit of normal; serum creatine<1.5-times upper limit of normal; PT≤upper limit of normal plus 6 seconds; INR≤2.3;
* sign up consent;
* unrolled by other clinical trials about hepatocellular carcinoma.

Exclusion Criteria:

* cannot tolerate TACE or TAI;
* CNS or bone metastasis exits;
* known history of other malignancy;
* be allergic to related drugs;
* underwent organ transplantation before;
* be treated before (interferon included);
* known history of HIV infection;
* known history of drug or alcohol abuse;
* have GI hemorrhage or cardiac/brain vascular events within 30 days;
* pregnancy;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
recurrence-free survival (RFS) | From date of randomization until the date of recurrence, assessed up to 60 months
  recurrence-free survival

SECONDARY OUTCOMES:
recurrence rate | 1 year, 2 year, 3 year, 5 year after surgery
  recurrence rate
Overall survival (OS) | From date of randomization until the date of death from any cause, assessed up to 60 months
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center of Sun Yat-Sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided